CLINICAL TRIAL: NCT00296166
Title: A Randomized Study That Will Show the Effects of Catheter Ablation Compared to the Effects of Thoracoscopic Ablation to Patients With Permanent Atrial Fibrillation.
Brief Title: Catheter Ablation Versus Thoracoscopic Ablation to Patients With Permanent Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients with permanent AF are seldomly symptomatic enough to justify intervention. We decided to stop inclusion due to low recruitment rate.
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAT-SKOPI study; KF - 01-284215
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2007-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Permanent Atrial fibrillation; catheter ablation; thoracoscopy; Arrhythmia; Heart
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Catheter ablation
Procedure: Thoracoscopic epicardial ablation

SUMMARY:
Patents with atrial fibrillation can be treated with the purpose of curing the arrhythmia.This may be achieved by catheter ablation and Maze surgery where the latter includes open heart surgery.

By catheter ablation the arrhythmia can be cured in about 70 % of patients who have episodes of atrial fibrillation. In patients with permanent atrial fibrillation the results are not as good.

We will compare a conventional ablation approach where lesions are created on the inside of the heart with a thoracoscopic approach where the lesions are created from the outside of the heart.

DETAILED DESCRIPTION:
Patients with permanent atrial fibrillation will be considered for randomisation Patients will be randomised to either conventional endocardial catheter ablation or epicardial thoracoscopic ablation.

Objectives of study:

Primary endpoint:presence of sinus rhythm after 6 months Secondary endpoints: complications, cost-effectiveness, structural changes (evaluated by echocardiography), p-BNP and inflammatory markers, atrial fibrillation burden evaluated by Holter monitoring

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrillation documented on at least 2 ecg´s with more than 1 month between ecg´s. The diagnosis is verified on Holter.
* All patients have symptoms or do not tolerate rate control treatment.

Exclusion Criteria:

* Psychiatric disease or suspicion of incapability to give informed concent
* Females with birth giving potential
* Previous heart surgery
* Previous ablation for atrial fibrillation
* Life expectance less than 1 year
* Congenital heart disease
* Expected need for heart surgery
* Heart failure (NYHA class IV)
* Inability to be treated with anticoagulation
* In case of previous deep venous thromboembolism og stroke the investigators will individually consider if the patient is suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-11; Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Presence of sinus rhythm | after 6 months from treatment

SECONDARY OUTCOMES:
complications | during 12 months from treatment
cost-effectiveness | during 12 months from treatment
structural changes (evaluated by echocardiography) | during 12 months from treatment
p-BNP | during 12 months from treatment
inflammatory markers | during 12 months from treatment
atrial fibrillation burden evaluated by Holter monitoring | at 6 months from treatment
exercise performance | at 3 months from treatment
Quality of life | at 3 months from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Svendsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Risghospitalet,, Copenhagen, Denmark